CLINICAL TRIAL: NCT00716300
Title: Functional Studies of High Density Lipoprotein in the Metabolic Syndrome
Brief Title: High Density Lipoprotein (HDL) Functionality in Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Western Australia (Other)
Responsible Party: Prof Gerald F Watts, University of Western Australia
Other Study IDs: DC-HDL2008
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Metabolic Syndrome X
Keywords: obesity; CVD; HDL kinetics; Anti-inflammatory and anti-oxidation studies; 30 subjects recruited (15 MetS and 15 lean controls)
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: obese and insulin resistant subjects
- 2: lean and normolipidaemic subjects

SUMMARY:
The aim of the study is to examine the kinetic, anti-oxidant, anti-inflammatory and cellular cholesterol efflux properties of high-density lipoprotein (HDL) in subjects with the metabolic syndrome (MetS) and lean individuals.

DETAILED DESCRIPTION:
Background and Purpose of This Study:

The metabolic syndrome (MetS) is characterized by impaired glucose and insulin metabolism (insulin resistance), abnormal body fat distribution called central obesity (a pot belly) and high blood pressure. People with the metabolic syndrome have markedly increased risk of heart disease which is mainly attributed to the abnormal fat metabolism and its associated metabolic disorders. Therefore, understanding of the body fat disorder is important to reduce the incidence and severity of heart disease.

Fats in the blood originate from dietary sources and from production by the liver. They are then delivered into peripheral body cell for utilization or storage. A particular protein, called high-density lipoprotein (HDL) apolipoprotein (apo) A-I, is an important fat carrier responsible for transporting excess fat from cells, via the bloodstream, back to the liver. Low HDL-apoA-I concentration is related to increased risk of heart disease. Subjects with MetS have reduced level of apoA-I and we wish to test the hypothesis that it is responsible for the impaired movement of fat from the periphery to the liver. Recent evidence suggests that the functionality of HDL, including anti-oxidant, anti-inflammatory and cholesterol efflux properties, is also important in preventing the development of heart disease. However, these function tests have not yet been investigated extensively in MetS.

Consequently, we wish to examine the transport and anti-atherogenic properties of HDL in subjects with MetS and compare these with normal lean subjects. Such findings would be of significant clinical importance in the understanding of the diverse role of HDL-apoA-I in reducing or preventing the progression of heart disease.

Participation:

Patients with MetS or lean individuals will be recruited for the study via newspaper advertisements. Following informed consent and once found suitable for participation, 15 men with MetS and 15 lean men will be enrolled. We will give the participants a harmless substance called a stable (non-radioactive) isotope. The isotope will trace the speed at which apoA-I is released into the blood (production) and are removed from the bloodstream (clearance) by the liver.

Participants will be asked to fast (only water allowed) for 12 hours prior to the isotope study. The stable isotope will be administered by intravenous injection in the form of a clear fluid (total volume approximates 15 to 25ml, 1-1.5 tablespoons). A small plastic tube (a cannula) will be placed into a vein in the arm, from where a total of 160mll (10.5 tablespoons) of blood will be obtained. The isotope study lasts 10 hours, during which participants will rest quietly and be allowed water only. At the end of the study day, participants will be given a meal and will be allowed home by taxi or family transport.

These studies will allow us to measure the metabolic action of apolipoprotein A-I, thereby gaining a better understanding of the mechanisms that leads to abnormal blood fat levels in those with MetS. To complete this study, each participant is required to attend 7 visits over a 6-week period.

Benefits:

All participants will receive health education, as well as information on personal health status and a review of heart risk factors.

ELIGIBILITY:
Inclusion Criteria:

MetS :the presence of at least three of the following:

* waist circumference > 102 cm, triglycerides > 1.7 mmol/L, HDL cholesterol < 1.05 mmol/L
* blood pressure ≥ 130/ ≥ 85 mmHg
* fasting glucose > 6.1 mmol/L

Lean control:

* BMI < 25 kg/m2
* waist circumference < 102 cm
* triglycerides < 1.0 mmol/L
* HDL-cholesterol > 1.3 mmol/L

Exclusion Criteria:

* subjects with plasma LDL-cholesterol > 5 mmo/L
* diabetes mellitus (defined by oral glucose tolerance test)
* genetic hyperlipidaemia (e.g. FH)
* consumption of > 30 g alcohol/day
* apolipoprotein E2/E2 genotype
* macroproteinuria
* creatinaemia ( > 120 umol/L)
* hypothyroidism
* hepatic dysfunction (AST or ALT > 2x ULN)
* major systemic illness and use of steroids or other agents that may influence lipid metabolism
* cardiovascular event within the past 6 months
* subjects on hypocaloric diets
* anaemia; any significant illness that in the opinion of reviewing physician would bear on the study (e.g. heart murmur or psychiatric conditions)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 men with features of the metabolic syndrome 15 age-matched normolipidaemic men
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald F Watts, MBBS, Principal Investigator — The University of Western Australia
Locations (1):
- University of Western Australia, Perth, Western Australia, Australia